CLINICAL TRIAL: NCT01470339
Title: Improvement the Anti-migraine Treatment Efficacy by Tailoring the Drug to Individual's Pain Modulation Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, d_yarnitsky, Professor, Head on Neurology Department, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 0462-10-RMB.CTIL
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Pain
Keywords: endogenous pain modulation; migraine; fMRI; duloxetine; preventive migraine treatment
MeSH Terms: conditions — Pain; Migraine Disorders | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): migraine patients to receive placebo treatment
  Interventions: Drug: duloxetine
- duloxetine (Active Comparator): migraine patients to receive duloxetine
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: duloxetine — duloxetine 60mg once a day for 5 weeks

SUMMARY:
* To delineate brain mechanisms that subserve endogenous analgesic (EA) in the healthy state.
* To identify alterations in mechanisms supporting EA in chronic pain (migraine) and their therapeutic relevance.

DETAILED DESCRIPTION:
The proposed research will use psychophysics and multiparametric MRI to (i) delineate the brain mechanisms that subserve and regulate endogenous analgesia (EA)in the healthy state and (ii) to identify alterations in mechanisms supporting EA in chronic pain and their therapeutic relevance. In both healthy subjects and chronic pain patients, EA will be probed using the DNIC (diffuse noxious inhibitory controls) and offset analgesia paradigms. Functional MRI will examine activation of brainstem mechanisms important in EA, while both functional and structural connectivity analyses will assess the regulation of these brainstem mechanisms by cerebral cortical regions involved in attention and affect. One pathological painful condition, migraine, will be examined since it allows changes in EA associated with chronic pain to be investigated between episodes of pain. Finally, EA and EA associated structural and functional parameters will be used to predict the efficacy of one compound, amitriptyline, to treat migraine in individual patients. Taken together, the proposed research will provide substantial insights into basic mechanisms supporting and regulating EA and can provide a foundation for mechanism-based individualized choice of therapy that may benefit all chronic pain patients.

ELIGIBILITY:
Inclusion Criteria:

* healthy females
* migaine females
* ages 18-50
* for migraineurs: >4 attacks/month

Exclusion Criteria:

* any migraine preventive treatment received during last 3 months or prior treatment with amytriptiline
* other chronic pain conditions
* psychiatric, other neurological diseases, language barrier or cognitive dysfunction
* Patients and controls will be asked to withdraw from any pain-relieving medications for 24 hours before the testing. The tests will be performed interictally atleast 2 days after the last attack.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2011-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Distinguish between two endogenous pain modulation mechanisms | 2 year

SECONDARY OUTCOMES:
To charcterize functional and structural neuroanatomical correlates of pain modulation profile and it's relevance for predicting the duloxetine efficacy in migraine | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David Yarnitsky, professor, Principal Investigator — Rambam Health Care Campus
Locations (1):
- MRI center, Haifa, Israel